CLINICAL TRIAL: NCT06347133
Title: Double-blind, Placebo-controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Plozasiran in Adults With Hypertriglyceridemia
Brief Title: Phase 3 Study of Plozasiran in Adults With Hypertriglyceridemia
Acronym: MUIR-3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AROAPOC3-3009; 2023-509302-30 (EudraCT Number)
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — plozasiran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plozasiran Injection (Experimental): 4 doses of plozasiran by subcutaneous (sc) injection
  Interventions: Drug: Plozasiran Injection
- Placebo (Placebo Comparator): calculated volume to match active treatment by sc injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Plozasiran Injection — ARO-APOC3 Injection
  Other Names: ARO-APOC3
  Arms: Plozasiran Injection
Drug: Placebo — sterile normal saline (0.9% NaCl)
  Arms: Placebo

SUMMARY:
This Phase 3 study will evaluate the safety and efficacy of plozasiran injection (ARO-APOC3) in adult participants with hypertriglyceridemia (HTG). After providing informed consent eligible participants will be randomized to receive 4 doses (once every 3 months) of plozasiran or placebo and be evaluated for efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Males, or nonpregnant (who do not plan to become pregnant) nonlactating females, who are ≥18 years of age at screening
* Established diagnosis of hypertriglyceridemia (HTG) and prior documented evidence (medical history) of mean fasting TG level ≥150 mg/dL (≥1.69 mm/L) and ≤499 mg/dL (≤5.64 mmol/L)
* Mean fasting TG level ≥150 mg/dL (≥1.69 mmol/L) and ≤499 mg/dL (≤5.64 mmol/L) collected at 2 separate and consecutive visits at least 7 days apart and no more than 17 days apart during the screening period
* Fasting low density lipoprotein-cholesterol (LDL-C) ≤ 130 mg/dL (≤3.37 mmol/L) at screening
* Screening HbA1c ≤9.0%
* Willing to follow diet counseling and maintain a stable low-fat diet
* Must be on standard of care lipid and TG-lowering medications per local guidelines (unless documented as intolerant as determined by the Investigator, including an inability to safely administer or re-administer a specific drug because of fear, preference, genetic, clinical, or metabolic considerations, or due a previous adverse reaction associated with, attributed to, or caused by specific drug) prior to collection of qualifying TG levels.

Exclusion Criteria:

* Use of any hepatocyte-targeted small interfering ribonucleic acid (siRNA) that targets lipids and/or triglycerides within 365 days before Day 1 (except inclisiran, which is permitted). Administration of investigational drug and inclisiran must be separated by at least 4 weeks.
* Use of any other hepatocyte targeted siRNA or antisense Oligonucleotide molecule within 60 days or within 5-half-lives before Day 1 based on plasma pharmacokinetics (PK), whichever is longer
* Acute pancreatitis within 4 weeks prior to screening
* Body mass index >45 kg/m^2

Note: Additional Inclusion/Exclusion criteria may apply per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1456 (Actual)
Dates: Start 2024-05-21 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Fasting Serum Triglyceride (TG) Levels from Baseline to Month 12 Compared to Placebo | Baseline, Month 12

SECONDARY OUTCOMES:
Percent Change in Fasting Serum TG Levels from Baseline to Month 10 Compared to Placebo | Baseline, Month 10
Proportion of Participants who Achieve Fasting TG Levels of <150 mg/dL (<1.69 mmol/L) at Month 12 Compared to Placebo | Month 12
Percent change in remnant cholesterol (VLDL-C) from baseline to Month 12 compared to placebo. | Baseline, Month 12
Percent change in non-HDL-C from baseline to Month 12 compared to placebo | Baseline, Month 12
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) Over Time through Month 12 as Compared to Placebo | From first dose of study drug through Month 12
Incidence Rates of New-Onset Diabetes Mellitus (NODM) Throughout the Course of Treatment | From first dose of study drug through Month 12
Incidence Rates of Impaired Glucose Tolerance Throughout the Course of Treatment | From first dose of study drug through Month 12
Incidence Rates of Worsening of Existing Diabetes Throughout the Course of Treatment | From first dose of study drug through Month 12
Change from Baseline in Hemoglobin A1c (HbA1c) and Other Glycemic Control Parameters During the Treatment Period Compared to Placebo | From first dose of study drug through Month 12
Change from Baseline in Fasting Blood Glucose During the Treatment Period Compared to Placebo | From first dose of study drug through Month 12
Change from Baseline in C-peptide During the Treatment Period Compared to Placebo | From first dose of study drug through Month 12
Change from Baseline in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) During the Treatment Period Compared to Placebo | From first dose of study drug through Month 12
Change from Baseline in Treatment-Emergent Adverse Events (TEAEs) and Treatment-Related Adverse Events (TRAEs) Associated with Worsening Glycemic Control During the Treatment Period Compared to Placebo | From first dose of study drug through Month 12
Initiation of New Medication for Hyperglycemia Among Study Participants Not Known to Have Pre-existing Diabetes Mellitus During the Treatment Period Compared to Placebo | From first dose of study drug through Month 12
Adjudicated Major Adverse Cardiovascular Events (MACE) Rates During the Treatment Period Compared to Placebo | From first dose of study drug through Month 12
Incidence of Anti-drug Antibodies (ADA) to Plozasiran in Participants Receiving Plozasiran Over Time Through Month 12 | From first dose of study drug through Month 12
Titers of Anti-drug Antibodies (ADA) to Plozasiran in Participants Receiving Plozasiran Over Time Through Month 12 | From first dose of study drug through Month 12

CONTACTS AND LOCATIONS:
Locations (235):
- United States (97):
  - Research Site 1, Birmingham, Alabama
  - Research Site 2, Mobile, Alabama
  - Research Site 3, Beverly Hills, California
  - Research Site 4, Canoga Park, California
  - Research Site 5, Garden Grove, California
  - Research Site 6, Huntington Beach, California
  - Research Site 7, Lake Forest, California
  - Research Site 8, Lincoln, California
  - Research Site 9, Long Beach, California
  - Research Site 10, Montclair, California
  - Research Site 11, Oxnard, California
  - Research Site 12, Redding, California
  - Research Site 13, Van Nuys, California
  - Research Site 14, Colorado Springs, Colorado
  - Research Site 15, Clearwater, Florida
  - Research Site 16, Hialeah, Florida
  - Research Site 17, Lake City, Florida
  - Research Site 18, Miami Lakes, Florida
  - Research Site 19, Mt. Dora, Florida
  - Research Site 20, North Miami Beach, Florida
  - Research Site 21, Orlando, Florida
  - Research Site 22, Pensacola, Florida
  - Research Site 23, Sarasota, Florida
  - Research Site 24, Tamarac, Florida
  - Research Site 25, Lawrenceville, Georgia
  - Research Site 26, Macon, Georgia
  - Research Site 27, Savannah, Georgia
  - Research Site 28, Sugar Hill, Georgia
  - Research Site 29, Park Ridge, Illinois
  - Research Site 30, Elkhart, Indiana
  - Research Site 31, Indianapolis, Indiana
  - Research Site 32, South Bend, Indiana
  - Research Site 33, Overland Park, Kansas
  - Research Site 34, Topeka, Kansas
  - Research Site 35, Louisville, Kentucky
  - Research Site 36, Zachary, Louisiana
  - Research Site 37, Annapolis, Maryland
  - Research Site 38, Baltimore, Maryland
  - Research Site 39, Flint, Michigan
  - Research Site 40, Minneapolis, Minnesota
  - Research Site 41, Olive Branch, Mississippi
  - Research Site 42, Jefferson City, Missouri
  - Research Site 43, St Louis, Missouri
  - Research Site 44, Norfolk, Nebraska
  - Research Site 46, Omaha, Nebraska
  - Research Site 45, Omaha, Nebraska
  - Research Site 47, Las Vegas, Nevada
  - Research Site 48, Summit, New Jersey
  - Research Site 52, New York, New York
  - Research Site 51, New York, New York
  - Research Site 53, Riverhead, New York
  - Research Site 54, Rochester, New York
  - Research Site 49, The Bronx, New York
  - Research Site 50, The Bronx, New York
  - Research Site 55, Vestal, New York
  - Research Site 56, Asheboro, North Carolina
  - Research Site 57, Morehead City, North Carolina
  - Research Site 58, Wilmington, North Carolina
  - Research Site 59, Winston-Salem, North Carolina
  - Research Site 60, Beavercreek, Ohio
  - Research Site 61, Cincinnati, Ohio
  - Research Site 63, Columbus, Ohio
  - Research Site 62, Columbus, Ohio
  - Research Site 64, Norman, Oklahoma
  - Research Site 66, Oklahoma City, Oklahoma
  - Research Site 65, Oklahoma City, Oklahoma
  - Research Site 67, Horsham, Pennsylvania
  - Research Site 68, Newport, Pennsylvania
  - Research Site 69, Newport, Pennsylvania
  - Research Site 70, Philadelphia, Pennsylvania
  - Research Site 71, Wilkes-Barre, Pennsylvania
  - Research Site 72, Fort Mill, South Carolina
  - Research Site 73, Greenville, South Carolina
  - Research Site 74, Chattanooga, Tennessee
  - Research Site 75, Powell, Tennessee
  - Research Site 76, El Paso, Texas
  - Research Site 77, Fort Worth, Texas
  - Research Site 86, Houston, Texas
  - Research Site 84, Houston, Texas
  - Research Site 85, Houston, Texas
  - Research Site 78, Houston, Texas
  - Research Site 80, Houston, Texas
  - Research Site 83, Houston, Texas
  - Research Site 82, Houston, Texas
  - Research Site 79, Houston, Texas
  - Research Site 81, Houston, Texas
  - Research Site 87, Laredo, Texas
  - Research Site 88, Missouri City, Texas
  - Research Site 89, Plano, Texas
  - Research Site 90, San Antonio, Texas
  - Research Site 91, Sugar Land, Texas
  - Research Site 92, Tomball, Texas
  - Research Site 93, Victoria, Texas
  - Research Site 94, Bountiful, Utah
  - Research Site 95, St. George, Utah
  - Research Site 96, Manassas, Virginia
  - Research Site 97, Seattle, Washington
- Argentina (9):
  - Research Site 102, CABA, Buenos Aires
  - Research Site 100, CABA, Buenos Aires
  - Research Site 103, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Research Site 104, Córdoba, Córdoba Province
  - Research Site 98, Córdoba, Córdoba Province
  - Research Site 101, Godoy Cruz, Mendoza Province
  - Research Site 105, Rosario, Santa Fe Province
  - Research Site 99, Rosario, Santa Fe Province
  - Research Site 106, Córdoba
- Australia (4):
  - Research Site 107, Blacktown, New South Wales
  - Research Site 108, Merewether, New South Wales
  - Research Site 110, Clayton, Victoria
  - Research Site 109, Heidelberg Heights, Victoria
- Bulgaria (27):
  - Research Site 111, Blagoevgrad
  - Research Site 112, Burgas
  - Research Site 113, Byala
  - Research Site 114, Dimitrovgrad
  - Research Site 115, Haskovo
  - Research Site 116, Kyustendil
  - Research Site 117, Pleven
  - Research Site 118, Pleven
  - Research Site 120, Plovdiv
  - Research Site 119, Plovdiv
  - Research Site 121, Plovdiv
  - Research Site 122, Rousse
  - Research Site 123, Sevlievo
  - Research Site 137, Sofia
  - Research Site 133, Sofia
  - Research Site 126, Sofia
  - Research Site 129, Sofia
  - Research Site 132, Sofia
  - Research Site 130, Sofia
  - Research Site 131, Sofia
  - Research Site 135, Sofia
  - Research Site 124, Sofia
  - Research Site 125, Sofia
  - Research Site 127, Sofia
  - Research Site 134, Sofia
  - Research Site 128, Sofia
  - Research Site 136, Stara Zagora
- Canada (12):
  - Research Site 140, North Vancouver, British Columbia
  - Research Site 141, Victoria, British Columbia
  - Research Site 142, Brampton, Ontario
  - Research Site 143, Sarnia, Ontario
  - Research Site 144, Waterloo, Ontario
  - Research Site 145, Chicoutimi, Quebec
  - Research Site 146, Laval, Quebec
  - Research Site 149, Montreal, Quebec
  - Research Site 139, Québec, Quebec
  - Research Site 147, Québec, Quebec
  - Research Site 148, Québec, Quebec
  - Research Site 138, Halifax
- Czechia (14):
  - Research Site 151, Prague, Prague
  - Research Site 157, Brno
  - Research Site 154, Hodonín
  - Research Site 159, Hradec Králové
  - Research Site 160, Náchod
  - Research Site 162, Olomouc
  - Research Site 155, Ostrava
  - Research Site 152, Prague
  - Research Site 156, Praha 4-Krc
  - Research Site 150, Slaný
  - Research Site 163, Teplice
  - Research Site 158, Trutnov
  - Research Site 161, Uherské Hradiště
  - Research Site 153, Ústí nad Labem
- France (4):
  - Research Site 164, Marseille, Bouches du Rhone
  - Research Site 167, Pessac, Gironde
  - Research Site 166, Lyon, Rhone
  - Research Site165, Paris
- Germany (3):
  - Research Site 170, Deggingen, Baden-Wurttemberg
  - Research Site 169, Wallerfing, Bavaria
  - Research Site 168, Magdeburg, Saxony-Anhalt
- Hungary (13):
  - Research Site 171, Békéscsaba
  - Research Site 175, Budapest
  - Research Site 183, Budapest
  - Research Site 179, Budapest
  - Research Site 184, Budapest
  - Research Site 180, Budapest
  - Research Site 182, Kaposvár
  - Research Site 176, Miskolc
  - Research Site 172, Pécs
  - Research Site 177, Pécs
  - Research Site 178, Szeged
  - Research Site 173, Veszprém
  - Research Site 174, Zalaegerszeg
- Italy (5):
  - Research Site 186, Rozzano, Milano
  - Research Site 187, Palermo, Sicily
  - Research Site 189, Bologna
  - Research Site 185, Brescia
  - Research Site 188, Milan
- Poland (19):
  - Research Site 200, Bydgoszcz
  - Research Site 202, Bydgoszcz
  - Research Site 192, Elblag
  - Research Site 193, Gdynia
  - Research Site 190, Katowice
  - Research Site 197, Krakow
  - Research Site 204, Krakow
  - Research Site 201, Lodz
  - Research Site 191, Lodz
  - Research Site 194, Malbork
  - Research Site 199, Szczecin
  - Research Site 207, Torun
  - Research Site 205, Warsaw
  - Research Site 198, Warsaw
  - Research Site 196, Wroclaw
  - Research Site 208, Wroclaw
  - Research Site 206, Wroclaw
  - Research Site 195, Zamość
  - Research Site 203, Żarów
- Slovakia (10):
  - Research Site 214, Banská Bystrica
  - Research Site 212, Bardejov
  - Research Site 217, Bratislava
  - Research Site 216, Bratislava
  - Research Site 210, Košice
  - Research Site 213, Moldava nad Bodvou
  - Research Site 209, Nové Zámky
  - Research Site 211, Prešov
  - Research Site 215, Rožňava
  - Research Site 218, Žilina
- South Africa (10):
  - Research Site 221, Centurion, Gauteng
  - Research Site 222, Krugersdorp, Gauteng
  - Research Site 228, Pretoria, Gauteng
  - Research Site 224, Durban, KwaZulu-Natal
  - Research Site 227, Cape Town, Western Cape
  - Research Site 219, Cape Town, Western Cape
  - Research Site 223, Cape Town, Western Cape
  - Research Site 225, Cape Town, Western Cape
  - Research Site 220, Somerset West, Western Cape
  - Research Site 226, Pretoria
- Spain (6):
  - Research Site 234, Barcelona, Barcelona
  - Research Site 229, A Coruña, La Coruña
  - Research Site 230, Barcelona
  - Research Site 232, Madrid
  - Research Site 231, Valencia
  - Research Site 233, Zaragoza
- United Kingdom (2):
  - Research Site 236, Plymouth, Devon
  - Research Site 235, London

IPD SHARING:
Plan to Share IPD: No